CLINICAL TRIAL: NCT03165916
Title: A Randomized Controlled Prospective Study to Compare the Incidence of Biliary Complications After Liver Transplantation
Brief Title: Study to Compare the Incidence of Biliary Complications After Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Scanga, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 140143
Record Dates: First submitted 2017-05-18; First posted 2017-05-24 (Actual); Results first posted 2020-07-30 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Liver Transplant; Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Reconstruction with stent placement (Experimental): Subjects will undergo biliary reconstruction with stent placement at the anastomosis site.
  Interventions: Device: Bard 5 Fr diameter feeding tube
- Reconstruction without stent placement (No Intervention): Subjects will undergo biliary reconstruction without stent placement.

INTERVENTIONS:
Device: Bard 5 Fr diameter feeding tube — A pediatric feeding tube is used as a stent over which biliary anastomosis is performed. This is not a permanent stent and generally migrates out on its own.
  Arms: Reconstruction with stent placement

SUMMARY:
A randomized prospective study will be conducted of patients at Vanderbilt University Medical Center who undergo liver transplantation from March 2014 until approximately 120 patients are randomized. Patients will be randomized to undergo biliary reconstruction with and without stent placement.

DETAILED DESCRIPTION:
The risk of biliary complications can be related to the type of liver transplant performed and the technique used for reconstruction of the bile duct. One of the main techniques of performing biliary reconstruction is a choledocholedochostomy which can be performed over an anastomotic stent. Although placement of biliary stents is routine practice in many liver transplant centers around the country, there is no clear evidence to support their use. As of now both the placement and non-placement of a stent are essentially "standard of care". In the investigators' center, many of the transplant surgeons now perform the biliary anastomosis over a pediatric feeding tube which is used as a stent. The practice of using stents in biliary anastomosis is not uniform and there are no established guidelines to support their indiscriminate application. The investigators have designed a prospective randomized trial to evaluate the effect of stent placement on biliary complications and its effect on morbidity.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* will be undergoing liver transplantation
* able to give informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Scanga, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Medical Center Liver Transplant Clinic, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 146 pts enrolled in study. 1 pt w/drew consent prior to randomization. 30 pts were inappropriate candidates & weren't randomized. 115 pts were randomized. 1 pt's clinical course required a second procedure & they were randomized twice. Initially the pt randomized to not receive a stent & later to receive a stent, there were 116 interventions.
Period: Overall Study
Arm/Group | Reconstruction With Stent Placement | Reconstruction Without Stent Placement
Started | 58 | 57
Reconstruction Interventions | 59 | 57
Completed | 58 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were 116 interventions but only 115 participants. A participant's clinical course necessitated a second procedure, and as such, they were randomized twice. The pt was initially randomized to not receive a stent and then randomized to receive a stent during the second procedure. Demographics are based on the first randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Reconstruction With Stent Placement | Reconstruction Without Stent Placement | Total
Number analyzed (Participants) | 58 | 57 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 33 | 71
  >=65 years | 20 | 24 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 15 | 38
  Male | 35 | 42 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 54 | 55 | 109
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 51 | 54 | 105
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 58 | 57 | 115

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biliary Complications
Description: Biliary complications include biliary strictures, biliary leaks, cholangitis, and stones. The investigators will compare the number of complications between the group that receives the stent and the group that does not.
Time Frame: 6 months after transplantation
Population: There was lack of significant difference between intervention groups so it was decided to not proceed with original 2 year analysis plan.
Measure: Number; unit: participants
Arm/Group | Reconstruction With Stent Placement | Reconstruction Without Stent Placement
Number analyzed (Participants) | 58 | 57
participants | 19 | 12

2. Primary Outcome: Number of Participants With Biliary Complications
Description: as for outcome 1
Time Frame: 12 months after transplantation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Reconstruction With Stent Placement | Reconstruction Without Stent Placement
Number analyzed (Participants) | 58 | 57
Participants | 19 | 14

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse event monitoring/assessing was limited to biliary complications related to procedure.
Arm/Group | Reconstruction With Stent Placement | Reconstruction Without Stent Placement
All-Cause Mortality (participants affected / at risk) | 2/58 | 7/57
Serious Adverse Events (participants affected / at risk) | 19/58 | 14/57
Other Adverse Events (participants affected / at risk) | 0/58 | 0/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reconstruction With Stent Placement (N=58) | Reconstruction Without Stent Placement (N=57)
Biliary Complications (Hepatobiliary disorders) | 19 (38) | 14 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-09-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT03165916/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT03165916/ICF_001.pdf